CLINICAL TRIAL: NCT05383300
Title: Investigating the Effect of Oxytocin and the Neurochemistry of Antisocial Personality Disorder and Psychopathy Using Neuroimaging
Brief Title: Intranasal Oxytocin in Antiosocial Personality Disorder and Psychopathy
Acronym: OXYASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Father Flanagan's Boys' Home (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 15/LO/1086
Record Dates: First submitted 2022-04-19; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2021-12

CONDITIONS: Antisocial Personality Disorder
Keywords: Oxytocin; Psychopathy; Violent Offenders; Social Processing
MeSH Terms: conditions — Antisocial Personality Disorder

STUDY DESIGN:
Intervention Model Description: Double-binded placebo-controlled crossover trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded- participant and investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Violent offenders with psychopathy (Other): Violent offenders with psychopathy
  Interventions: Drug: Oxytocin nasal spray; Other: Placebo spray
- Violent offenders without psychopathy (Other): Violent offenders without psychopathy
  Interventions: Drug: Oxytocin nasal spray; Other: Placebo spray
- Healthy non-offenders (Other): Healthy non-offenders
  Interventions: Drug: Oxytocin nasal spray; Other: Placebo spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal spray containing 40 IU of oxytocin
Other: Placebo spray — Application of inert placebo, identical in odor, color, and droplet size except for absence of oxytocin

SUMMARY:
A pharmacoimaging study of oxytcoin in antisocial personality disorder and psychopathy

DETAILED DESCRIPTION:
Using a double-blinded, placebo controlled design, we explored similarities and differences in i) an important component of empathic processing (neural response to facial emotional expressions) and ii) decision-making in violent men with ASPD+/-Psychopathy, compared to healthy non-offenders (NO; n= 21 across studies), with placebo and after acute application of intranasal oxytocin, using functional Magnetic Resonance Imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-60
* IQ greater than 70 as defined by the Wechsler Abbreviated Scale of Intelligence (WASI-II).

Violent offenders:

Offenders with convictions for violent crimes (murder, rape, attempted murder, grievous and actual bodily harm) who met DSM-5 criteria for antisocial personality disorder (Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5 PD) Psychopathy or non-psychopathy subgroup based on Psychopathy Checklist- Revised (PCL-R; (Hare, 2003))- score of 25 as the threshold for psychopathy in this English population.

Healthy non-offenders:

Non-offenders with no personality disorder

Exclusion criteria:

* history of major mental disorders (bipolar 1, bipolar 2, major depression or psychotic disorders)
* self-reported neurological disorders
* head injury resulting in loss of consciousness for 1 hour or longer
* severe visual or hearing impairments
* contraindications to MRI

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Within-group effect of oxytocin on nerual modulation of fear | 10 minutes
  Differences in responsivity to morphed faces on FMRI in oxytocin vs fear condition- clusterwise analysis using AFNI (effect size is beta values)

SECONDARY OUTCOMES:
Baseline neural modulation of morphed fearful faces | 10 minutes
  Response to morphred faces on FMRI in placebo condition- clusterwise analysis using AFNI (effect size is beta values)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Blackwood, MB MD, Principal Investigator — King's College London
Locations (1):
- Insititue of Psychiarty, Psychology and Neuroscience, London, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This was not built into original ethical protocol due to concerns about sensitivity of data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT05383300/Prot_SAP_000.pdf